CLINICAL TRIAL: NCT06522061
Title: Evaluating the Effective and Safe Use of Stream™ Platform by a Lay User in a Simulated Environment
Brief Title: Evaluating the Effective and Safe Use of Stream™ Platform
Acronym: Home-Stream
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FluidAI Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLS0009
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: User-Centered Design; Anastomotic Leak; Colorectal Surgery; Artificial Intelligence
Keywords: Anastomotic Leak; Artificial Intelligence; Colorectal Surgery; ERAS; Stream Platform
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Masking Description: The investigators, care providers, participants, and outcome assessors will be blinded to the anastomotic leak risk-score generated by Stream Platform. This will ensure that subject care is not influenced by use of the device and postoperative monitoring is conducted as per the standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Arm (Experimental): Stream™ Platform will be attached to the abdominal/pelvic drains of the patients enrolled in this group. The platform will conduct continuous pH and electrical conductivity measurements of the abdominal drain fluid.
  All subjects recruited will take part in the evaluation of Stream™ Platform in a simulated home-use environment.
  Interventions: Device: Stream™ Platform

INTERVENTIONS:
Device: Stream™ Platform — Stream™ Platform consists of 5 main components: Origin™, Delta™ Monitor, Stream™ Application, Accessory Calibration Syringe(s), and Stream™ Cart. Origin™ is an inline biosensor system that can be attached between an off-the-shelf drainage catheter and evacuator bag/bulb system and is designed to monitor real-time changes in drained effluent characteristics (specifically pH and electrical conductivity (EC)) for the early identification of postoperative complications. Origin™ requires daily calibration (via Accessory Calibration Syringe(s)) for optimal performance and accuracy of its sensors. The Stream Application is a mobile application for displaying and analyzing data collected continuously via Origin™. Stream™ Application is pre-installed on Android mobile devices (called Delta™ Monitor) that are supplied by FluidAI. Origin connects to Stream Application via Bluetooth. Mobile carts/mounts, denoted Stream™ Carts/Delta Mounts, will be used to house the Delta™ Monitor.

SUMMARY:
The study aims to demonstrate the potential for at-home monitoring using Stream™ Platform, through simulated-use testing. Lay users, defined as subjects or nonprofessional caregivers, will be asked to operate Stream™ Platform. Safety, efficacy, and usability data will be collected to ensure that users are able to comply with prescribed device use.

Additionally, clinical testing will be conducted to identify correlations between measurements from Stream™ Platform and standard laboratory, radiological, and clinical assessments used for leak detection as part of the current standard of care (SOC) that may be skipped if the subject is discharged early.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years - male or female.
* Subject/SDM understands and has voluntarily signed and dated Informed Consent Form (ICF).
* Subject underwent colorectal surgery with anastomosis.
* Subjects must be willing to comply with trial requirements.
* Subject has a prophylactic abdominal/pelvic drain after colorectal surgery.

Exclusion Criteria:

* Subjects/caregiver is unwilling or unable to comply with the requirements of the protocol.
* 24 hours or more have passed since the end of the subject's surgery and consent was not attained.
* The subject had already developed an anastomotic leak at the time of screening and underwent surgery for treatment of the complication.
* Plans that the subject will be discharged in less than 3 days post-surgery.
* Subject has reported that they are pregnant.
* Subject has a permanent end stoma.
* Subject is delirious.
* Subject has severe dementia.
* Subject was involved in the planning and conduct of the clinical investigation.
* Origin™ is not compatible with the drain used on the subject.
* Subject and/or caregiver is/are not capable of conducting the calibrations for Stream™ Platform (this can be self-reported or determined by the CRC/HCP/other research staff).
* The subject and/or caregiver is/are unable to understand the instructions provided for the management and calibration of Stream™ Platform (this can be self-reported or determined by the CRC/investigator/other research staff).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate if lay users can operate Stream Platform safely and effectively under healthcare providers supervision (simulated home use) | Through study completion, an average of 6-months
  1. Statistical evaluation of the number of calibration errors encountered due to lay user error as reported by the healthcare providers.
  2. Statistical evaluation of the number of calibration errors due to lay user errors that required intervention by the supervising healthcare provider to protect subject health and safety.
  3. Occurrence of device associated adverse events including:
  i. Adverse Device Events (ADE) ii. Serious Adverse Device Events (SADE) iii. Unanticipated Serious Adverse Device Events (USADE) iv. Device Deficiencies
Evaluate lay users' satisfaction through user feedback survey | Through study completion, an average of 6-months
  Subject reported overall satisfaction with daily calibrations and overall device.
  The following parameters will be recorded on a scale of 1-5:
  1. System Related Feedback
     * Overall feedback on Stream Platform
     * Overall feedback on Stream Application
  2. Training Related Feedback
     * Overall feedback on the instructions provided by Stream Application
     * Overall feedback on the training material provided including but not limited to training video, infographic, etc.
     * Overall feedback on the in-person training conducted
  3. Subject Comfort Assessment
     * Overall subject experience performing ADLs (Activities of Daily Living) while Stream Platform is in use.
     * Overall subject experience sleeping while Stream Platform is in use

SECONDARY OUTCOMES:
Utilize continuous pH and EC measurements collected prospectively using Stream™ Platform to supplement FluidAI's existing clinical model for early prediction of leakage after colorectal surgery. | Through study completion, an average of 6-months
  Data collected will be used to supplement Stream™ Platform's existing clinical model for early prediction of leakage.
Identify correlations between measurements from Stream™ Platform and current standard of care (SOC). | Through study completion, an average of 6-months
  Assess if any strong correlations exist between pH/EC measurement collected using FluidAI's Stream™ Platform and other diagnostic biomarkers for AL
Estimate the time taken by lay users to conduct calibration procedures | Through study completion, an average of 6-months
  Quantify the average time taken by subjects/caregiver to conduct calibration in seconds as measured by the Stream™ Platform

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul's Hospital - Providence Healthcare (PHC), Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No